CLINICAL TRIAL: NCT05244161
Title: Effectiveness of Early Child Development Multi-Media Communication on Caregiver and Community Health Worker Behaviors: Evaluation of the Malezi II Program
Brief Title: A Quasi-experimental Evaluation of the Malezi Program in Tanzania
Acronym: Malezi II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Ministry of Health, Community Development, Gender, Elderly and Children (Unknown); President's Office, Regional Administration and Local Government (Unknown); Development Media International (Other); Aga Khan University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EG0227
Record Dates: First submitted 2022-01-25; First posted 2022-02-17 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Child Development; Father-Child Relations; Knowledge, Attitudes, Practice; Safety Issues
Keywords: Early child development; Parenting; Media intervention; Community health workers; Program evaluation; Caregiver
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radio messaging (RM) (No Intervention): Radio messaging only (RM)
- RM, Video job aids, Early Childhood Development program (RMV-ECD) (Active Comparator): Radio messaging, short video job aids primarily for CHW use, and the UNICEF Care for Childhood Development program (RMV-ECD)
  Interventions: Behavioral: RMV-ECD

INTERVENTIONS:
Behavioral: RMV-ECD — Combined radio messaging, video job aids (primarily for CHWs), Care for Childhood Development package
  Arms: RM, Video job aids, Early Childhood Development program (RMV-ECD)

SUMMARY:
The quality of caregiving and the parent-child relationship is critical for early child development (ECD) and has been shown to be modifiable. This study evaluated an ECD project in Tanzania, assessing the effectiveness of radio messaging (RM) alone and a combined radio messaging/video job aids/ECD (RMV-ECD) intervention, using a two-arm pre-post design study, which enrolled a cohort of caregivers of children 0-24 months in four districts of Tabora region, following them for nine months. ECD radio messages were broadcast on popular stations at least 10 times/day reaching all study districts. In two districts, community health workers (CHW) trained in UNICEF's Care for Child Development package and used ECD videos in home- and facility-based sessions with caregivers. Five outcomes were used to assess the intervention effects: ECD knowledge, early stimulation, father engagement, responsive care, and environment safety. Additionally the effect of the training and video job aids on the quality of CHWs' counseling support was evaluated primarily using structured observation checklists of household visits and facility group counseling sessions with caregivers and their children. Qualitative data was collected from a subset of caregivers and CHW participating in the study to assess acceptability and other perceptions of the project.

DETAILED DESCRIPTION:
Standardized interventions aimed at supporting child development are successful in a variety of cultural and socio-economic contexts, particularly in low to middle income countries. Integrated community and facility-based interventions can improve parenting behaviors. Mass media radio messaging campaigns can increase caregiver and community knowledge, and caregiver motivation to seek appropriate health care through reaching a broader audience such as family/household influencers such as fathers or grandparents.

Study design and setting:

This was a two-arm quasi-experimental pre-post evaluation study, comparing different 9-month intervention packages to establish their relative impact on parenting skills and environment among a cohort of caregivers of children under age three years in Tabora region, located in central-western Tanzania and home to a predominantly rural (87%) population. The study included four districts divided into two intervention groups. The first group (Kaliua, Uyui districts) was exposed to the minimal intervention package, composed of radio messaging (RM) only. The second group (Nzega, Igunga districts) was exposed to the Malezi II full intervention package, composed of radio messaging, the introduction of short video job aids primarily for community health worker (CHW) use, and the UNICEF Care for Childhood Development (CCD) program (RMV-ECD).

Sample and sampling procedures:

As the comprehensive program intervention was primarily delivered by CHW who were affiliated with health facilities, 31 health facilities were purposefully selected located in 29 administrative units called wards (6-8/district). From these wards, 75 National Bureau of Statistics census enumeration areas (EA) were randomly sampled proportional to population size. The study team aimed to enumerate all households in sampled EAs, listing potentially eligible households if there was a resident adult (>18 years) primary caregiver of a child aged 0-24 months who intended to remain in the same area for at least one year, and was willing to be home-visited by a CHW. From these listed households, only one caregiver per household was recruited. Caregivers who were not able to provide written informed consent due to a cognitive impairment or language barrier; or who were the primary caregiver of an index child with a congenital anomaly or other disability; or who worked as a CHW or medical provider, were excluded from the study.

The study team estimated that a completed sample size of 430 caregivers per intervention group would provide 90% power to detect a 15% difference between the RM and RMV-ECD intervention groups at endline, and >80% power to detect at least a 5% change in each t intervention group between baseline and endline, at a 5% significance level. Of 8880 households enumerated, 1248 caregivers were recruited into the study and interviewed at baseline (October-December 2019). Of these, 1051 were eligible for follow-up; 1004 (96%) were successfully traced and interviewed at endline (January-March 2021). Almost all (n=985; 98%) caregivers interviewed at endline remained the primary caregiver of the index child from baseline. Of the 19 caregivers whose index child had died or moved from the household, eight nominated an eligible "replacement" child under three years and 11 completed a partial interview skipping questions that were no longer applicable.

A cohort of 120 CHWs was also enrolled from the two intervention districts, who were assigned to caregiver-cohort enrolled households in the RMV-ECD arm.

Data collection and study variables Structured questionnaires were administered in a private place in or near the consenting caregiver's home in the national language (Swahili). Five outcome variables were defined reflecting caregiver knowledge, stimulation practices, father engagement, responsive care, and household environment risk. Continuous scores for each variable were dichotomized at the median for analysis. Some scores, where the number of items differed by age of the child (early stimulation) or sub-group (environment risk), were standardized to a 0-1 scale by dividing the raw score by the number of items. The quality of CHWs counseling support was evaluated using a structured evaluation checklist, targeting two home and two clinic observations for each CHW in each round; pre and post intervention. The checklist had 23 items across 6 dimensions; introduce, educate, ask, plan/problem solve, interact/encourage, and responsive care. Under the qualitative process evaluation, 25 in-depth interviews (IDI) were completed with caregivers enrolled in the cohort, and four focus group discussions (FGD) were held among those in the CHW cohort.

ELIGIBILITY:
Households who had:

Inclusion Criteria:

* resident adult (>18 years) primary caregiver of a child aged 0-24 months, and had the
* intention to remain in the same area for at least one year,
* willingness to be home-visited by a Community Health Worker.

Exclusion Criteria:

* unable or unwilling to give informed consent

CHW eligibility criteria:

* assigned to a Malezi II study health facility/catchment community
* working as a Malezi II project CHW (i.e. attended Malezi (I or II) training, or capacitated for Malezi II project through on-job training and mentoring)
* able to understand and willing to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1248 (Actual)
Dates: Start 2019-10-13 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Caregiver age appropriate early childhood development knowledge as assessed by responses to interview-administered questions | 9 months
  Proportion of respondents scoring <2 (poor knowledge) or 2-6 (good knowledge) to six questions (scoring 0-6 points) asking the caregiver to describe one specific way that a "caregiver can support a child's mental, emotional or physical development…" during pregnancy, from birth to six months, from 6-9, 9-12, and 12-24 months and 2-5 years of age. Caregiver responses coded correct or incorrect.
Caregiver early childhood stimulation practices as assessed by responses to interview-administered questions adapted from UNICEF's Multiple Indicator Cluster Surveys | 9 months
  Proportion of respondents scoring poor (<50%) or good (equal or >50%) to questions on stimulation. Caregivers of children under seven months could score up to three points for reporting that the mother, father, or other adult engaged the child in singing songs, taking the child outside, or playing with the child in the past week. Caregivers of children over seven months were asked three additional items (read books, told stories, name/count things with child) for a total of six points. The sum of the items for these two measures were then standardized to a 0-1 scale.
Father engagement with the child as assessed by caregiver responses to interview-administered questions adapted from UNICEF's Multiple Indicator Cluster Surveys | 9 months
  Proportion of respondents scoring <2 (poor engagement) or 2-6 (good engagement) to questions on father engagement. Caregivers of children under seven months could score up to three points for reporting that the father engaged the child in singing songs, taking the child outside, or playing with the child in the past week. Caregivers of children over seven months were asked three additional items (read books, told stories, name/count things with child) for a total of six points. The sum of the items for these two measures were then standardized to a 0-1 scale.
Responsive care as assessed by interviewer observations of how the caregiver engaged with the child during the interview using questions from the interview guide | 9 months
  Proportion of respondents scoring <5 (poor responsive care) or 5-6 (good responsive care) by observed by interviewers of how the caregiver engaged with the child during the interview. Observations consisted of four items totaling up to six points which included helping the child keep busy (0, 1), pointing out objects/naming things (scored as 0, 1), recognizing when the child needs help with something (0,1,2), and keeping the child in view at all times (0,1,2).
Household environment risk as assessed by interviewer observation of the inner and outer household areas using questions from interview guide | 9 months
  Proportion of respondent households scoring equal or <0.3 (poor) or >0.3 (good) to interviewer observations of household and neighborhood environment safety from risks of community (nearby road, bar/market, ditches); outside compound (open water source, unpenned animals, accessible sharp tools, chemicals or flammable materials, and unprotected cooking area); and inside household (accessible electric, medicine or cleaning chemicals, inappropriate toys). The environment risk outcome was standardized (0-1) to adjust for the different number of items in each group.
Quality of CHWs counseling assessed by independent observations of home and clinic counseling sessions against a checklist | 12-18 months
  Proportion of CHWs scoring <15 or (poor) equal or >16 (good) on quality of home and clinic counseling at baseline and endline from video observations based on a 23-item checklist assessing how CHW 1) introduce topic/session, 2) educate on appropriate activities, 3) ask caregivers about behaviors, 4) plan and problem-solve, 5) interact with and encourage caregivers, and 6) discuss responsive care. Items with yes" or "no" response options were scored as "1" or "0", and items with "well done," "partly" or "not done" responses were scored "1," "0.5" or "0" points, respectively. Raw scores were then standardized to a 0-1 scale. Clinic and home observations scored separately and subsequently combined for an overall score.

SECONDARY OUTCOMES:
Acceptability of ECD intervention activities as assessed through open-ended responses recorded in in-depth interviews with caregivers and focus group discussions with CHW. | 9-12 months
  Among CHW, perceptions and experiences receiving project training and implementing ECD intervention activities (home visits, videos, group counseling, radio). Among caregivers, perceptions and experiences of CHW support and receiving the ECD intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Elizabeth Glaser Pediatric AIDS Foundation, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antelman G, Ferla J, Gill MM, Hoffman HJ, Komba T, Abubakar A, Remes P, Jahanpour O, Mariki M, Mang'enya MA, van de Ven R. Effectiveness of an integrated multilevel early child development intervention on caregiver knowledge and behavior: a quasi-experimental evaluation of the Malezi program in Tanzania. BMC Public Health. 2023 Jan 4;23(1):19. doi: 10.1186/s12889-022-14956-2. PMID 36600280

DOCUMENTS (1):
  • Study Protocol (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT05244161/Prot_000.pdf